CLINICAL TRIAL: NCT04202341
Title: Long-Term, Observational, Global Registry of Patients With Generalized Myasthenia Gravis Who Have Received Treatment With Complement C5 Inhibition Therapies (C5ITs)
Brief Title: Registry of Participants With Generalized Myasthenia Gravis Treated With Alexion C5 Inhibition Therapies (C5ITs)
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALXN-MG-501
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis
Keywords: gMG; Soliris; Ultomiris; Alexion C5 Inhibition Therapy; Alexion C5IT; Patient Registry; Generalized Myasthenia Gravis; Alexion Registry
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term, multicenter, multinational, observational, registry of patients with gMG that is designed to collect data on clinical outcomes and safety in patients prescribed Alexion C5 inhibitor therapies (C5IT) such as eculizumab (Soliris®) and ravulizumab (Ultomiris®).

DETAILED DESCRIPTION:
At the time of enrollment in the Registry, participant records will be queried for retrospective information about the participants' medical history and gMG disease treatment history. Following enrollment, prospective data collection will be performed using data obtained as part of the routine clinical care and through patient-reported outcome methods in use. Data will be collected using an electronic data capture system. The duration of data collection for the Registry will be up to 5 years from the day of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a diagnosis of gMG who are treated with Alexion C5IT at the time of enrollment, including patients previously treated with Soliris or Ultomiris and withdrawn from treatment.
2. Capable of giving signed informed consent, which includes compliance with the protocol requirements and restrictions.
3. Participants must have myasthenia gravis historical data, such as MG-ADL and MGFA class, available to be enrolled in the Registry.

Exclusion Criteria:

1. Participants currently enrolled in an Alexion-sponsored interventional clinical study for treatment of gMG cannot be enrolled in the Alexion gMG Registry while enrolled/participating in the clinical study for gMG therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of gMG who are treated with Alexion C5IT at the time of enrollment, or have ever been treated with Alexion C5IT prior to enrollment, and meet the inclusion criteria and exclusion criteria are eligible for registry participation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Myasthenia Gravis Activities of Daily Living (MG-ADL) Score | Approximately 5 years from enrollment
  The MG-ADL is an eight-item patient-reported outcome measure assessing MG symptoms and functional activities related to activities of daily living.48 Each of the items is scored from 0 (normal) to 3 (most severe), providing a total MG-ADL score ranging from 0 to 24, where higher scores indicate greater severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (32):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Scottsdale, Arizona
  - Clinical Trial Site, Fresno, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, Rancho Mirage, California
  - Clinical Trial Site, Sylmar, California
  - Clinical Trial Site, Colorado Springs, Colorado
  - Clinical Trial Site, Fort Collins, Colorado
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Clearwater, Florida
  - Clincal Trial Site, Gainesville, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Augusta, Georgia
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Lexington, Kentucky
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Lansing, Michigan
  - Clinical Trial Site, Columbia, Missouri
  - Clinical Trial Site, New Hyde Park, New York
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Dayton, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Chattanooga, Tennessee
  - Clinical Trial Site, Knoxville, Tennessee
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Burlington, Vermont
  - Clinical Trial Site, Milwaukee, Wisconsin
- Clinical Trial Site, Vienna, Austria
- Canada (3):
  - Clinical Trial Site, Brampton, Ontario
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Montreal, Quebec
- China (9):
  - Clinical Trial Site, Chengdu, Sichuan
  - Clinical Trial Site, Beijing
  - Clinical Trial Site, Changchun
  - Clinical Trial Site, Chengdu
  - Clinical Trial Site, Guangzhou
  - Clinical Trial Site, Jinan
  - Clinical Trial Site, Nanchang
  - Clinical Trial Site, Qingdao
  - Clinical Trial Site, Shijiazhuang
- Clinical Trial Site, Hanover, Hannover, Germany
- Italy (2):
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Naples
- Saudi Arabia (3):
  - Clinical Trial Site, Abhā
  - Clinical Trial Site, Jeddah
  - Clinical Trial Site, Riyadh